CLINICAL TRIAL: NCT04301063
Title: An International Multicentric Open-label Descriptive Study to Assess the Effects and Evaluate the Tolerance of the Cosmetic Care Product RV3278A in the Follow-up Phase of Facial Acne in Teenagers and Young Adults for 1 Year
Brief Title: Assess the Effects and the Tolerance of Cosmetic Product in the Follow-up Phase of Facial Acne for 1 Year
Status: Completed | Type: Observational
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Other Study IDs: RV3278A2018244
Record Dates: First submitted 2019-11-14; First posted 2020-03-09 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-04

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Cyanoacrylate skin surface stripping (CSSS) of the stratum corneum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RV3278A arm: study product RV3278A is applied twice a day on the face during the whole study.
  In case of reaction resulting from the use of the product, the subject will inform the investigator who will explain to him/her what to do : application reduction or stop applications for a while
  Interventions: Other: RV3278A

INTERVENTIONS:
Other: RV3278A — RV3278A is a non-rinsed cosmetic cream intended to be used every day on adolescents and young adults with acne-prone skin.

SUMMARY:
Acne is a chronic inflammatory disease of the pilo-sebaceous unit in the skin. Indeed, your skin is covered with tiny holes called hair follicles, or pores. These pores contain sebaceous glands (also called oil glands) that make sebum, an oil that moistens your hair and skin. Most of the time, the glands make the right amount of sebum and the pores are fine. But sometimes a pore gets clogged up with too much sebum, dead skin cells, and germs called bacteria. This can cause acne.

Pierre Fabre Laboratories have developed a cosmetic care product, a cream which is commercialized since September 2019. This leave-on skin care product is adapted for acne-prone skin.

In this study, we are interested in the effects of this care product in facial acne evolution for 12 months (quality of life, acne severity, number of acne flares). Also, we are interested in the subject's satisfaction regarding the use of this care product. This study will also enable to know if the product is well tolerated in such application circumstances.

This clinical study will be carried out in 54 subjects (female or male), aged between 12 and 35 years, in about 10 centers in different European countries.

The maximal duration of the study for a subject will be 1 year. If you give your consent to take part in this study, you will receive a cosmetic care product, also called study product, that you will apply on your face twice a day (morning and evening) for the whole duration of the study.

What makes this study original is the use of a smartphone application to help you to comply with the study procedures and to help the investigator to follow you.

DETAILED DESCRIPTION:
Acne vulgaris is one of the most common skin conditions in teenagers that often persists into adulthood. It is a chronic inflammatory disease of the pilosebaceous unit resulting from four main factors: increase of sebum production, follicular hyperproliferation and hyperkeratinisation leading to comedones formation, inflammation and proliferation of the bacteria Propionibacterium acnes.1,2 Acne affects nearly all people between the ages of 15 and 17 years and in 15 to 20% of young people, acne is moderate to severe. The prevalence of acne in 12-24 years is 85%. 3 The presence of acne may have psychologic or emotional impact: it may negatively affect mood, quality of life and self-esteem in adolescents and adults and can increase the risk of anxiety, depression and suicidal ideation2,3. There is not always a correlation between the acne clinical severity and the quality of life.

According to its severity, the acne vulgaris can be treated locally with topical agents used alone or in combination, such as benzoyl peroxide, retinoids (adapalene…), antibiotics, azelaic acid, etc.

Oral treatments are usually taken for more severe acne and include antibiotics, contraceptives and isotretinoin. They also can be used in combination with local treatments.1,4

The product RV3278A is a non-rinsed cosmetic cream intended to be used every day on adolescents and young adults with acne-prone skin.

In accordance with the Pierre Fabre laboratories safety charter, a full program of tolerance has been performed including pre-clinical and clinical studies in healthy volunteers. The product presents a sufficient safety level to be used for this protocol.

The use of cosmetics in acne is well established. The goals of cosmetics in acne are

* to complement drug therapy, by alleviating their side effects and thereby improving treatment adherence.
* to contribute to improving the status of the clinically non-lesional skin.

Clinically non-lesional skin in acne patients (CNLSAP) is well known for its greasiness, which is due to overproduction of sebum.

Another important character of the CNLSAP is the "invisible microcomedone" (IMC).

1. IMC can be visualized by "stripping-it-out" with cyanoacrylate.
2. IMC is composed as a mixture of cellular components of the follicular infundibulum, and sebum lipids, both of which can be analysed ex-vivo by all tools of currently available technology.
3. IMC is considered to be the root of any subsequent clinical lesion, both non- inflammatory ones (open and close comedones microcysts) and inflammatory ones (papules pustules etc..)5
4. The number/cm2 and size of the IMC are highly variable and correlate with subsequent acne severity.
5. Therefore, any cosmetic product able to modify the number/cm2 and size of the IMC would contribute to maintain healthier skin in acne patients and reduce the use of drug therapy.

A pilot study in acne patients has shown that an herbal extract used topically for several weeks months was able to reach such goals.

The present study is aimed at reproducing these results in several dermatology practices in Europe.

ELIGIBILITY:
Inclusion Criteria:

Criteria related to the population:

* Female or male aged between 12 and 35 years included
* Phototype I, II, III or IV according to Fitzpatrick classification
* For major subject:

  o Subject who has signed his/her written informed consent for his/her participation in the study
* For minor subject:

  o Subject and/or parent(s)/legal representative(s), according to national regulations, who have signed his/her written informed consent for subject's participation in the study
* If required by national regulations, subject must be registered with health social security or health social insurance
* Woman of childbearing potential:

  o use of an effective contraceptive method, as assessed by the investigator, for at least 3 months before the inclusion, accepting to go on using this method during the whole duration of the study
* Subject or parent (s) / guardian(s) owning a smartphone with adequate parameters to download the application (including having enough storage space, a version of android or iOS compatible with the application) and a web access

Related to the diseases and skin condition:

* Subject with oily skin
* Subject with dilated pores on the forehead
* Almost clear, mild or moderate facial acne with score index severity GEA=1 (almost clear), GEA=2 (mild) or GEA=3 (moderate) assessed on a scale ranged from 0 to 5.

Exclusion Criteria:

Related to the population:

* Subject who is unable to understand the information given including study procedures (for linguistic or psychiatric reasons) and to give his/ her consent to participate
* Subject who is currently participating, plans to participate or has participated in another clinical study prior to inclusion visit, liable to interfere with the study assessments according to the investigator
* For woman of childbearing potential: subject pregnant or breastfeeding or planning to be pregnant during the study
* Subject deprived of freedom by administrative or legal decision or under guardianship
* Subject who, in the judgement of the investigator, is not likely to be compliant with study-related requirements
* Subject who is a family member of the investigator or any associate, colleague, employee assisting in the conduct of the study ( secretary, nurse, technician…)

Related to the disease:

* Severe type of acne (Acne conglobata, Acne fulminans or nodulocystic acne) or acneiform induced eruptions according to investigator's assessment
* Facial skin pathology other than acne, skin abnormalities or dermatological condition on the face liable to interfere with the study assessments (including psoriasis, atopic dermatitis, skin infectious disease of viral, bacterial, fungus or parasitic origin …)
* Forehead scars in tested area liable to interfere with samples realisation (cyanoacrylate stripping)
* Acute, chronic or progressive disease or medical history considered by the investigator hazardous for the subject or incompatible with the study or liable to interfere with the study assessments
* Clinical signs of hormonal dysfunctions or hyperandrogenism
* History of allergy or intolerance to any cosmetic product, to the investigational product ingredients or to cyanoacrylate
* Solar erythema on the face due to excessive UV exposure

Related to the treatments/products:

* Any surgery, chemical or physical treatment on the experimental area done within 6 months before the inclusion or planned during the study
* Oral intake of isotretinoin within 6 months before the inclusion
* Hormonal contraception or hormonal antic-acne treatment established or modified within 3 months before the inclusion or planned to be established or modified during the study
* Any oral or topical anti-acne treatment taken/applied on the face within 1 month before the inclusion
* Use of topical or systemic treatment during the previous weeks or ongoing, liable to interfere with the assessment of the cutaneous tolerance and effects of the studied product (according to the investigator's appreciation)
* Facial cleansing or skin care product containing anti-acne or keratolytic ingredients applied within 15 days before the inclusion or planned to be applied during the study
* Facial cleansing or skin care product (including moisturizer, make-up remover, foundation cream/powder) established or modified within 15 days before the inclusion
* Any rinsed/non-rinsed skin care product (including moisturizer and sunscreen), make-up (including foundation cream/powder) or make-up remover applied on the face (including eyes and mouth) the day of the inclusion visit

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects will be enrolled from the investigator's outpatients' reception. Subjects corresponding to eligibility criteria will be contacted by the investigator who will propose them to take part in the clinical study.
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2020-05-06 (Actual); Study Completion 2020-05-06 (Actual)

PRIMARY OUTCOMES:
Change in acne severity from Baseline to 365 days | Day 1, Day 35, Day 120, Day 180, Day 270, Day 365
  Global Evaluation Acne (GEA), a 6-point scale 0 : Clear, No lesions
  1. : Almost clear, Almost no lesions
  2. : Mild
  3. : Moderate
  4. Severe
  5. : Very severe
Number of acne relapse(s)/flare(s) | 1 year-period
  Acne flare or relapse are defined by the necessity to introduce an oral and/or facial anti-acne treatment and GEA score ≥3.
Change in Acne lesions counting | Day 1, Day 35, Day 120, Day 180, Day 270, Day 365
  Each type of acne lesions (non-inflammatory and inflammatory: open comedones, closed comedones, papules, pustules and nodules) will be counted on the whole face at each visit by the investigator according to the Lucky method
Change in Cardiff Acne Disability Index questionnaire (CADI) | Day 1, Day 180, Day 365
  It consists in 5 questions regarding the way the subject feels about the acne, each response is on a 4-point scale. The score is calculated by summing the score of each question resulting in a possible maximum of 15 and a minimum of 0. The higher the score, the more the quality of life is impaired.
Change in Subject's Global Assessment (SGA) of acne severity | Day 35, Day 120, Day 180, Day 270, Day 365
  The subject will assess the global severity of his/her acne on a 7-point scale in comparison to acne severity at baseline (visit 1):
  (-3) Very much worse (-2) Much worse (-1) Minimally worse (0) No change
  1. Minimally improved
  2. Much improved
  3. Very much improved
Change in pilosebaceous follicles status on forehead area | Day 1, Day 180 and Day 365 for the majority of the centres. 2 designated centres will performed it also at Day 35, Day 120 and Day 270
  Ex vivo analysis of pilosebaceous follicles will be performed by cyanoacrylate skin surface stripping method
Occurrence of Adverse events | 1 year
  It will be determined by the subject's / parent(s) or guardian(s) spontaneous reporting, the investigator's non-leading questioning, his/her critical review of the e-diary and his/her clinical evaluation
Change in Local tolerance | Day 1, Day 35, Day 120, Day 180, Day 270, Day 365
  by the Investigator using a 4-point scale for each physical or functional sign on the whole face: none, mild, moderate, severe
Change in Tolerance | Day 1, Day 35, Day 120, Day 180, Day 270, Day 365
  The following 5-point scale will be used by the investigator:
  * (1) Excellent: no functional nor physical signs related to the investigational product observed or reported by the subjects
  * (2) Very good
  * (3) Good
  * (4) Moderate
  * (5) Bad
Global Tolerance | Day 365
  Based on the same 5-point scale. The investigator will consider:
  * The type of reaction (discomfort, irritation, delayed/immediate allergic reaction) and its intensity, duration, recurrence, time of emergence
  * The population (age, acne skin…)
  * The type of product
Change in the subject statisfaction regarding the use of RV3278A | Day 1, Day 120, Day 365
  Questionnaire

CONTACTS AND LOCATIONS:
Locations (6):
- France (3):
  - Centre de Santé Sabouraud - Hôpital Saint Louis, Paris
  - cabinet Médical, Sèvres
  - Skin Research Centre, Toulouse
- Italy (2):
  - Medical Office, Milan
  - Medical Office, Pavia
- Medical Office, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No